CLINICAL TRIAL: NCT01366027
Title: PRISM Registry: Pseudobulbar Affect Registry Series
Status: Completed | Type: Observational
Sponsor: Avanir Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 11-AVR-REG-001
Record Dates: First submitted 2011-06-02; First posted 2011-06-03 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-04

CONDITIONS: Alzheimer's Disease; Amyotrophic Lateral Sclerosis (ALS); Multiple Sclerosis (MS); Parkinson's Disease; Stroke; Traumatic Brain Injury
Keywords: pseudobulbar affect
MeSH Terms: conditions — Alzheimer Disease; Amyotrophic Lateral Sclerosis; Multiple Sclerosis; Parkinson Disease; Stroke; Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
PBA is a neurologic condition that is estimated to impact over a million patients and their families in the United States. PBA occurs secondary to an otherwise unrelated neurologic disease or injury, and manifests as involuntary, frequent, and disruptive outbursts of crying and/or laughing. Progress has been made in better understanding this debilitating condition, but much more needs to be done. That's why a new PBA patient registry, PRISM (Pseudobulbar Affect RegIstry Series), has been initiated.

The goal of PRISM is to establish the prevalence and quality of life (QOL) impact of PBA in patients with underlying neurologic conditions including

* Alzheimer's disease
* Amyotrophic lateral sclerosis
* Multiple sclerosis
* Parkinson's disease
* Stroke
* Traumatic brain injury

Because this is an observational registry, it doesn't require you to intervene with any specific treatment or procedure. Your participation allows the PRISM registry to collect and analyze data from your site and also compare it to national numbers captured in the PRISM registry about PBA across all of the major at-risk neurologic populations.

ELIGIBILITY:
Inclusion Criteria:

* All participants must have underlying neurologic conditions known to be risk factors of PBA: Alzheimer's Disease, Amyotrophic Lateral Sclerosis, Multiple Sclerosis, Parkinson's Disease, Stroke, and Traumatic Brain Injury.
* The population for this study will be 18 years and over

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population for this study will be 18 years and over
Sampling Method: Probability Sample
Enrollment: 5290 (Actual)
Dates: Start 2011-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Prevalence of PBA (using CNS-LS) | Upon Study Enrollment/Entry
  The objective of the registry is to determine the prevalence of pseudobulbar affect (PBA) in patients with certain underlying neurologic conditions: Alzheimer's Disease (AD), Amyotrophic Lateral Sclerosis (ALS), Multiple Sclerosis (MS), Parkinson's Disease (PD), Stroke (STR), and Traumatic Brain Injury (TBI). Presence of PBA symptoms was defined as CNS-LS score >=13.

CONTACTS AND LOCATIONS:
Overall Officials: Randall Kaye, MD, Study Chair — Avanir Pharmaceuticals
Locations (1):
- Avanir Pharmaceuticals, Aliso Viejo, California, United States